CLINICAL TRIAL: NCT03738501
Title: Slow Expiratory Technique Efficacy on 24 Hours Food Ingestion in Children Under Than 12 Months, Hospitalized for Bronchiolitis : a Randomized Controlled Study
Brief Title: Slow Expiratory Technique to Improve Alimentation in Children With Bronchiolitis
Acronym: BRONCHIOL-EAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Principal Investigator, Yann Combret, Physiotherapist, MSc, PhD Candidate, Groupe Hospitalier du Havre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-A01864-51
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Acute Viral Bronchiolitis
Keywords: Food intake; Chest physiotherapy; Sleep; Respiratory Distress
MeSH Terms: conditions — Dyspnea | interventions — SET protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chest physiotherapy with SET (Experimental): Chest physiotherapy will be provided by a single physiotherapist not involved in outcomes assessment. Airway clearance technique will be Slow Expiratory Technique (SET). SET is a slow modulation of airflow in order to remove bronchial secretions within infants lungs. Experimental group will also benefit for standard medical and non-pharmacological care (e.g Standard Treatment)
  Interventions: Other: Chest physiotherapy with SET; Other: Standard Treatment
- Standard treatment (Active Comparator): Medical treatment, health education for parents, rhinopharyngeal clearance using isotonic saline solution, advices.
  Interventions: Other: Standard Treatment

INTERVENTIONS:
Other: Chest physiotherapy with SET — Chest physiotherapy with SET, and standard treatment (medical treatment, health education, nasopharyngeal clearance, advice)
  Arms: Chest physiotherapy with SET
Other: Standard Treatment — Standard pharmacological and non-pharmacological treatments (medical treatment, health education, rhinopharyngeal clearance, advices)

SUMMARY:
The purpose of this study is to determine wether a single chest physiotherapy session with slow expiratory technique (SET) improves infants with viral bronchiolitis quality of life (food intake and sleep) on the next 24 hours.

DETAILED DESCRIPTION:
Bronchiolitis is the most common lower respiratory viral infection in infants. Nowadays bronchiolitis is the first reason of children hospitalisation worldwide. Symptoms are based on airway inflammation associated to an increased mucus production and cell necrosis leading to a multifactorial airway obstruction. Recommended treatments are supportive care based on oxygenation and rehydration. Airway clearance techniques represented by chest physiotherapy remain controversial.

Considering that bronchiolitis impacts respiratory condition in young infants feeding and sleep may be reduced. Evaluating quality of life represented by feeding and sleep in hospitalized infants may be an important outcome in this population.

The investigators hypothesized that chest physiotherapy with SET will improve children's quality of life, especially 24 hours food intake and sleep.

ELIGIBILITY:
Inclusion Criteria:

* children under 12 months
* hospitalized for bronchiolitis
* chest physiotherapy prescription
* bronchial obstruction confirmed by physician and respiratory physiotherapist

Non-inclusion Criteria :

* children more than 1 year
* exclusive breastfeeding or enteral feeding
* prematurity (gestational age < 35 weeks)
* cardiac, neurological and pulmonary comorbidity
* continuous oxygen supplementation or ventilatory support
* chest physiotherapy contraindications

Exclusion Criteria:

* side effects during chest physiotherapy : bradycardia <100 bpm, oxygen saturation<90%, general state alteration
* outing, oxygen supplementation or parenteral nutrition less than 24 hours after randomization
* chest physiotherapy cessation according to family request

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Food ingestion | 24 hours following intervention
  Total Food ingestion within 24 hours after intervention measured by nurses or parents

SECONDARY OUTCOMES:
Sleep quality | 24 hours following intervention
  Total Sleep Time
Sleep quality | 24 hours following intervention
  Desaturation<90% (Pulse oximetry monitoring during sleep) count during diurnal and nocturnal sleep
Oxygen saturation | Before intervention ; 5 minutes, 30 minutes and 24 hours after intervention
  Pulse oximetry monitoring
Respiratory rate | Before intervention ; 5 minutes, 30 minutes and 24 hours after intervention
  Pulse oximetry monitoring
Heart Rate | Before intervention ; 5 minutes, 30 minutes and 24 hours after intervention
  Pulse oximetry monitoring
Respiratory Distress | Before intervention ; 5 minutes, 30 minutes and 24 hours after intervention
  Bronchiolitis Severity Score (described by Gajdos et al. as mentioned in the references). The Bronchiolitis Severity Score involves the calculation and addition of three subscores (age-based respiratory rate scale, score of 1-3; retractions, and wheeze scales, both running from 0 to 3). Total score ranges from 1 to 9, with higher scores indicating greater respiratory distress.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Le Roux, MD, Principal Investigator — Groupe Hospitalier du Havre
Locations (1):
- Groupe Hospitalier Du Havre, Le Havre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ralston SL, Lieberthal AS, Meissner HC, Alverson BK, Baley JE, Gadomski AM, Johnson DW, Light MJ, Maraqa NF, Mendonca EA, Phelan KJ, Zorc JJ, Stanko-Lopp D, Brown MA, Nathanson I, Rosenblum E, Sayles S 3rd, Hernandez-Cancio S; American Academy of Pediatrics. Clinical practice guideline: the diagnosis, management, and prevention of bronchiolitis. Pediatrics. 2014 Nov;134(5):e1474-502. doi: 10.1542/peds.2014-2742. PMID 25349312
- [Background] Gajdos V, Katsahian S, Beydon N, Abadie V, de Pontual L, Larrar S, Epaud R, Chevallier B, Bailleux S, Mollet-Boudjemline A, Bouyer J, Chevret S, Labrune P. Effectiveness of chest physiotherapy in infants hospitalized with acute bronchiolitis: a multicenter, randomized, controlled trial. PLoS Med. 2010 Sep 28;7(9):e1000345. doi: 10.1371/journal.pmed.1000345. PMID 20927359
- [Background] Gajdos V, Beydon N, Bommenel L, Pellegrino B, de Pontual L, Bailleux S, Labrune P, Bouyer J. Inter-observer agreement between physicians, nurses, and respiratory therapists for respiratory clinical evaluation in bronchiolitis. Pediatr Pulmonol. 2009 Aug;44(8):754-62. doi: 10.1002/ppul.21016. PMID 19598273
- [Derived] Combret Y, Machefert M, Couet M, Bonnevie T, Gravier FE, Gillot T, Le Roux P, Hilfiker R, Medrinal C, Prieur G. Effect of a prolonged slow expiration technique on 24-h food intake in children hospitalized for moderate bronchiolitis: a randomized controlled trial. Ital J Pediatr. 2024 Sep 27;50(1):196. doi: 10.1186/s13052-024-01770-2. PMID 39334411
- [Derived] Roque-Figuls M, Gine-Garriga M, Granados Rugeles C, Perrotta C, Vilaro J. Chest physiotherapy for acute bronchiolitis in paediatric patients between 0 and 24 months old. Cochrane Database Syst Rev. 2023 Apr 3;4(4):CD004873. doi: 10.1002/14651858.CD004873.pub6. PMID 37010196